CLINICAL TRIAL: NCT06691139
Title: A Comparative Study of Temporalis Fascia Graft and Periosteal Graft in Myringoplasty
Status: Completed | Type: Observational
Sponsor: Mohamed Soltan Nada (Other)
Responsible Party: Sponsor-Investigator, Mohamed Soltan Nada, Resident, otorhinolaryngology Head and neck department sohag university, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-med-15-10-11MS
Record Dates: First submitted 2024-11-01; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Myringoplasty
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Retrospective study, charts will be reviewed for 80 patients ages from 12 years to 40 years with complete records who underwent myringoplasty by otorhinolaryngologist at sohag university hospital from January 2022 to January 2024
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group (A) patients with periosteal graft: patients whose underwent to myringoplasty using periosteal graft
  Interventions: Procedure: Myringoplasty using periosteal graft and myringoplasty using Temporalis fascia graft in patients ages from 12 years to 40 years; Other: Myringoplasty using Temporalis fascia graft and myringoplasty using periosteal graft; Procedure: Myringoplasty operation using periosteal graft and myringoplasty using Temporalis fascia graft; Procedure: Group (A) myringoplasty using periosteal graft Group (B) Myringoplasty using Temporalis fascia graft
- (B) patients with Temporalis fascia graft: patients whose underwent to myringoplasty using Temporalis fascia graft
  Interventions: Procedure: Myringoplasty using periosteal graft and myringoplasty using Temporalis fascia graft in patients ages from 12 years to 40 years; Other: Myringoplasty using Temporalis fascia graft and myringoplasty using periosteal graft; Procedure: Myringoplasty operation using periosteal graft and myringoplasty using Temporalis fascia graft; Procedure: Group (A) myringoplasty using periosteal graft Group (B) Myringoplasty using Temporalis fascia graft

INTERVENTIONS:
Procedure: Myringoplasty using periosteal graft and myringoplasty using Temporalis fascia graft in patients ages from 12 years to 40 years — Myringoplasty using periosteal graft and myringoplasty using Temporalis fascia
Other: Myringoplasty using Temporalis fascia graft and myringoplasty using periosteal graft — Group (A) Myringoplasty using periosteal graft Group (B) Myringoplasty using Temporalis fascia graft
Procedure: Myringoplasty operation using periosteal graft and myringoplasty using Temporalis fascia graft — Myringoplasty using Temporalis fascia graft and myringoplasty using periosteal graft in age from 12years to 40 years
Procedure: Group (A) myringoplasty using periosteal graft Group (B) Myringoplasty using Temporalis fascia graft — Myringoplasty operation using Temporalis fascia graft and Myringoplasty using periosteal graft in patients from 12 years to 40 years

SUMMARY:
A Comparative Study of Temporalis Fascia Graft and Periosteal Graft in Myringoplasty

DETAILED DESCRIPTION:
The aim of this clinical trials is to asses and compare the surgical outcomes of Temporalis fascia graft and periosteal graft in myringoplasty in terms of graft intake and audiological improvement

ELIGIBILITY:
Inclusion Criteria:

age 12years to 40 years Small to moderate sized perforation . Dry tubotympanic chronic suppurative otitis media For more than 6 weeks .

Exclusion Criteria:

Active discharge or superimposed otomycosis . Patients with sensorineural hearing loss. Patients with considerable nasal pathology.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Sohag university hospital
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
hearing improvment | from January 2022 to January 2024
  outcome of temporalis fascia graft and periosteal graft for managment tympanic membrane perforation for audiological improvement

CONTACTS AND LOCATIONS:
Overall Officials: ahmed Nada, Principal Investigator — Sohag University
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No